CLINICAL TRIAL: NCT05311644
Title: La désensibilisation Aux Venins d'hyménoptères : Quelle Est Son efficacité à Long Terme ? (EFLOTITA2)
Brief Title: Hymenoptera Venom Immunotherapy: Evaluation of Its Long-term Efficacy at the University Hospital of Angers (EFLOTITA2)
Acronym: EFLOTITA2
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC20_0158
Record Dates: First submitted 2022-01-31; First posted 2022-04-05 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Anaphylaxis Caused by Hymenoptera Venom (Disorder)
Keywords: hymenoptera venom immunotherapy; anaphylaxis; venom allergy
MeSH Terms: conditions — Anaphylaxis; Venom Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Included: All participants that cesed VIT between 2005 and 2019, and did not withdraw his consent to participate to the study.
  Interventions: Other: Telephone survey

INTERVENTIONS:
Other: Telephone survey — All participants are interviewed by telephone, and are asked to answer a survey.

SUMMARY:
Allergy to Hymenoptera venom is one of the main causes of anaphylaxis in adults, and is less common in the paediatric population. It can be severe or even fatal.

Despite the use of an emergency kit, including an adrenaline auto-injector (AAI), at present only hymenoptera venom immunotherapy (VIT) is effective in preventing subsequent severe systemic reactions.

Recurrence during the 5 years following cessation of VIT is about 10-15 percent. Studies evaluating longer-term efficacy are scarce.

At the University Hospital of Angers, hundreds of patients are treated each year, and its allergology unit has been providing VIT for over 15 years.

The purpose of this stufy is to evaluate VIT efficacy among patients who were treated with VIT and ceased VIT from 2005 to 2019, at the university hospital of Angers.

DETAILED DESCRIPTION:
Allergy to Hymenoptera venom is one of the main causes of anaphylaxis in adults, and is less common in the paediatric population. It can be severe or even fatal.

Despite the use of an emergency kit, including an adrenaline auto-injector (AAI), at present only hymenoptera venom immunotherapy (VIT) is effective in preventing subsequent severe systemic reactions.

Recurrence during the 5 years following cessation of VIT is about 10-15 percent. Studies evaluating longer-term efficacy are scarce.

At the University Hospital of Angers, hundreds of patients are treated each year, and its allergology unit has been providing VIT for over 15 years.

The purpose of this stufy is to evaluate VIT efficacy among patients who were treated with VIT and ceased VIT from 2005 to 2019, at the university hospital of Angers.

This is a monocentric and ambispective study. In the absence of opposition from the patient (within one month after the information letter was sent), the search for data of interest is carried out by consulting the participant's medical record. An investigator (doctor or intern) interviews the participant, or the legal guardian for minors, and performs a telephone survey.

Data are collected from the participants medical records. Information gathered are as follows : age, sexe, the date and symptoms following hyménoptera stings, the evolution of allergy skin testing, total and venom specific immunoglobuin E (IgE), venom specifc immunoglobulin G4 (IgG4), basophil activation tests (BAT) to hymenoptera venom, exposure to hymenoptera stings.

The telephone survey assesses potential new comorbidities and new treatments, exposure to hymeoptera stings, hymenoptera stings after VIT cessation, if known : the hymenoptera specy, the participants reaction to the sting, and the drug that has been used to treat the symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Allergy to hymenoptera venom.
* Treated with VIT at the university hospital of Angers.
* Ceased VIT between 2005 and 2019.

Exclusion Criteria:

* Patient's opposition, or the Participant's legal guardian's, if minor, to participate to the study, and/or for his data to be used.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Allergy to hymenoptera venom, Treated with VIT at the university hospital of Angers, Ceased VIT between 2005 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Reccurence of a systemic reaction | up to 17 years since the patient ceased hymenoptera venom immunotherapy.
  The recurrence of a systemic reaction after a hymenoptera sting reported by the patient during the telephone survey.

SECONDARY OUTCOMES:
To describe the evolution of the results of the allergy work-up during hymenoptera venom immunotherapy | up to 17 years since the patient ceased hymenoptera venom immunotherapy to the last appointement in the allergy unit.
  Results of skin-testing and blood work
Predicting the recurrence of systemic symptoms | up to 17 years since the patient ceased hymenoptera venom immunotherapy until the phone survey
  To identify any predictor of the recurrence of systemic symptoms after discontinuation of hymenoptera venom immunotherapy, among the above listed parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Angers, Angers, Maine et Loire, France

IPD SHARING:
Plan to Share IPD: No